CLINICAL TRIAL: NCT00845871
Title: A Single-arm, Open-label Study of the Palatability and Tolerability of Deferasirox Taken With Meals, With Different Liquids or Crushed and Added to Food
Brief Title: Palatability and Tolerability of Deferasirox Taken With Meals, With Different Liquids or Crushed and Added to Food
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS32; 2011-004217-17 (EudraCT Number)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Transfusional Hemosiderosis
Keywords: Exjade; deferasirox; palatability; tolerability; food; iron overload; Serum Iron overload due to transfusions
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): Participants were administered daily with deferasirox starting dose of 20 mg/kg orally to a maximum dose of 40 mg/kg/day.
  Interventions: Drug: deferasirox:

INTERVENTIONS:
Drug: deferasirox: — Participants were administered daily with deferasirox starting dose of 20 mg/kg orally to a maximum dose of 40 mg/kg/day.
  Other Names: Exjade; Deferasirox

SUMMARY:
This single-arm, open-label, multi-center study enrolled 65 patients from approximately 20 centers. All patients who met the study criteria and were taking, beginning or resuming treatment with Deferasirox were allowed. The study will began with a one month run-in phase, where all patients were instructed to take Deferasirox according to their physician's prescribing information.

DETAILED DESCRIPTION:
Following the run-in phase, patients entered a three month, assessment phase. During the assessment phase, patients were given five general options for taking Deferasirox including with or without meals, crushed and added to a soft food or mixed in a liquid of choice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with thalassemia major, sickle cell disease (SCD), low or intermediate 1 (INT 1) risk myelodysplastic syndrome (MDS) or other anemias and transfusional hemosiderosis.
* Patients who were on, starting, or resuming treatment with Exjade.
* Patients who were >2 years (i.e., 2 years of age or older).

Exclusion criteria:

* Serum creatinine above the upper limit of normal (ULN) for age.
* Alanine aminotransferase (ALT) >2.5 times the ULN.-High risk intermediate-2 or high risk MDS or acute leukemia.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Children's Hospital and Research Center, Oakland, California
  - Stanford University, Palo Alto, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - University of Colorado Denver, Colorado Sickle Cell Treatment and Research Center, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Children's Hospital of Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - St Joseph Children's Hospital, Paterson, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Presbyterian Hospital, New York, New York
  - New York Medical College, Valhalla, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - St Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center and Hematology Services, Houston, Texas

REFERENCES:
- [Derived] Goldberg SL, Giardina PJ, Chirnomas D, Esposito J, Paley C, Vichinsky E. The palatability and tolerability of deferasirox taken with different beverages or foods. Pediatr Blood Cancer. 2013 Sep;60(9):1507-12. doi: 10.1002/pbc.24561. Epub 2013 Apr 23. PMID 23637051
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 centres in United States.
Pre-assignment Details: 82 participants were screened, out of which 65 participants enrolled into study. Study design comprised of a one-month run-in period where participants took deferasirox according to the physician, followed by a three-month assessment period. In assessment period, participants were instructed to document the selected method of administration and meal (breakfast, dinner, or no meal). Method of administration and meal type were kept same over week, but allowed to change once a new week began.
Groups:
- Deferasirox: Participants were administered with deferasirox starting dose of 20 milligram/kilogram/day (mg/kg/day), daily 30 minutes before meal for 4 weeks of Run-in period. Where as, Participants were administered daily with deferasirox at a minimum starting dose of 20 mg/kg/day along with different food and liquids consistently for 12 weeks of assessment period. For participants receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
Period: Run-in Period
Arm/Group | Deferasirox
Started | 65
Completed | 65
Not Completed | 0
Period: Assessment Period
Arm/Group | Deferasirox
Started | 65
Completed | 58
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Abnormal laboratory values | 1
Not completed — Abnormal test procedure results | 1
Not completed — Patient withdrew consent | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed in Intent-to-treat (ITT) population defined as all enrolled patients regardless of any treatment received or not. As per the planned analysis, data was summarized as overall by combining all Arms/Groups.
Groups:
- Deferasirox: Participants were administered daily with deferasirox at a minimum starting dose of 20 mg/kg/day along with different food and liquids consistently for 12 weeks of assessment period. For participants receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
Arm/Group | Deferasirox
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (22.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 26
  Black | 25
  Asian | 10
  Other | 4
Taking Exjade prior to the study [Count of Participants; unit: Participants]
  Yes | 44
  No | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Differing Palatability Scores at Week 8 and Week 12
Description: Palatability was assessed by participants based on a five-point Facial Hedonic scale defined as: dislike extremely; somewhat dislike; neither like or dislike; somewhat like; like extremely for the meal and method of administration. For participants under 5 years of age, the scale was completed by parent or caregiver.
Time Frame: Week 8 and Week 12
Population: The primary analysis was performed in the ITT population defined as all subjects enrolled regardless of any treatment received or not. As per the planned analysis, data were summarized by counts and percentages of each category of response when administered with food or with different methods of administration.
Measure: Number; unit: percentage of participants
Groups:
- Breakfast (Deferasirox With Soft Food): Participants received crushed deferasirox at a minimum starting dose of 20 mg/kg/day added to soft food at breakfast for 12 weeks of assessment period. For participants receiving > 30 mg/kg/ day, a maximum of 40 mg/kg/day was allowed.
- Breakfast (Deferasirox With Liquid): Participants received deferasirox at a minimum starting dose of 20 mg/kg/day dispersed in a beverage of choice (non-carbonated, non-alcoholic liquid) at breakfast for 12 weeks of assessment period. For participants receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
- Dinner (Deferasirox With Soft Food): Participants received crushed deferasirox at a minimum starting dose of 20 mg/kg/day added to soft food a dinner for 12 weeks of assessment period. For participants receiving > 30 mg/kg/ day, a maximum of 40 mg/kg/day was allowed.
- Dinner (Deferasirox With Liquid): Participants received deferasirox at a minimum starting dose of 20 mg/kg/day dispersed in a beverage of choice (non-carbonated, non-alcoholic liquid) at dinner for 12 weeks of assessment period. For participants receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
- No Meal (Deferasirox With Liquid): Participants received deferasirox at a minimum starting dose of 20 mg/kg/day dispersed in a beverage of choice (non-carbonated, non-alcoholic liquid) with no meal for 12 weeks of assessment period. For participants receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
- No Meal Deferasirox With Soft Food): Participants received crushed deferasirox at a minimum starting dose of 20 mg/kg/day added to a soft food with no meal for 12 weeks of assessment period. For participants receiving > 30 mg/kg/ day, a maximum of 40 mg/kg/day was allowed.
Arm/Group | Breakfast (Deferasirox With Soft Food) | Breakfast (Deferasirox With Liquid) | Dinner (Deferasirox With Soft Food) | Dinner (Deferasirox With Liquid) | No Meal (Deferasirox With Liquid) | No Meal Deferasirox With Soft Food)
Number analyzed (Participants) | 16 | 11 | 6 | 10 | 40 | 17
percentage of participants
  Week 8, Dislike extremely: number analyzed (Participants) | 10 | 7 | 3 | 7 | 17 | 7
  Week 8, Dislike extremely | 10 | 0 | 0 | 0 | 0 | 0
  Week 8, Somewhat dislike: number analyzed (Participants) | 10 | 7 | 3 | 7 | 17 | 7
  Week 8, Somewhat dislike | 0 | 28.6 | 0 | 14.3 | 5.9 | 14.3
  Week 8, Neither like or dislike: number analyzed (Participants) | 10 | 7 | 3 | 7 | 17 | 7
  Week 8, Neither like or dislike | 20 | 28.6 | 33.3 | 28.6 | 29.4 | 28.6
  Week 8, Somewhat like: number analyzed (Participants) | 10 | 7 | 3 | 7 | 17 | 7
  Week 8, Somewhat like | 30 | 0 | 0 | 28.6 | 17.6 | 42.9
  Week 8, Like extremely: number analyzed (Participants) | 10 | 7 | 3 | 7 | 17 | 7
  Week 8, Like extremely | 40 | 42.9 | 66.7 | 28.6 | 47.1 | 14.3
  Week 12, Dislike extremely: number analyzed (Participants) | 6 | 4 | 3 | 3 | 23 | 10
  Week 12, Dislike extremely | 0 | 0 | 0 | 0 | 4.3 | 0
  Week 12, Somewhat dislike: number analyzed (Participants) | 6 | 4 | 3 | 3 | 23 | 10
  Week 12, Somewhat dislike | 0 | 25 | 0 | 0 | 4.3 | 10
  Week 12, Neither like or dislike: number analyzed (Participants) | 6 | 4 | 3 | 3 | 23 | 10
  Week 12, Neither like or dislike | 16.7 | 25 | 0 | 33.3 | 56.5 | 50
  Week 12, Somewhat like: number analyzed (Participants) | 6 | 4 | 3 | 3 | 23 | 10
  Week 12, Somewhat like | 33.3 | 0 | 66.7 | 33.3 | 8.7 | 10
  Week 12, Like extremely: number analyzed (Participants) | 6 | 4 | 3 | 3 | 23 | 10
  Week 12, Like extremely | 50 | 50 | 33.3 | 33.3 | 26.1 | 30

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuation and Interruption
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards. Subjects who had permanently terminated from the treatment or kept the treatment on hold/deviated from protocol due to adverse event were defined as subjects with permanent discontinuation and temporary interruption, respectively.
Time Frame: Day 1 up to Week 16
Population: The analysis was performed in the Safety Set (SAF) population, defined as all participants who received at least one dose of study medication. As per the planned analysis, data were summarized by counts and percentages of each category of response when administered with food or with different methods of administration.
Measure: Count of Participants; unit: Participants
Groups:
- Deferasirox (Run-in Phase): Participants were administered with deferasirox starting dose of 20 milligram/kilogram/day (mg/kg/day), daily 30 minutes before meal.
Arm/Group | Deferasirox (Run-in Phase) | Breakfast (Deferasirox With Soft Food) | Breakfast (Deferasirox With Liquid) | Dinner (Deferasirox With Soft Food) | Dinner (Deferasirox With Liquid) | No Meal (Deferasirox With Liquid) | No Meal Deferasirox With Soft Food)
Number analyzed (Participants) | 62 | 20 | 18 | 14 | 17 | 39 | 30
Participants
  AEs | 39 | 10 | 6 | 6 | 6 | 24 | 11
  SAEs | 5 | 5 | 0 | 1 | 1 | 6 | 0
  AEs leading to permanent discontinuation | 0 | 2 | 0 | 0 | 0 | 0 | 1
  AEs leading to temporary interruption | 4 | 2 | 1 | 0 | 0 | 2 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Trough Plasma Concentration of Deferasirox at Week 8, Week 12 and Week 16
Description: Blood samples were drawn at every visit as close as possible to 24 hours post dose from each subject participating in the study and trough plasma concentrations were estimated.
Time Frame: Pre-dose (0), 1, 2, 4 and 6 hour (post-dose) at Week 8, 12 and 16
Population: The analysis was performed in the ITT population defined as all subjects enrolled regardless of any treatment received or not. As per the planned analysis, data was summarized as overall by combining all Arms/Groups.
Measure: Median (Full Range); unit: micromoles per litre (μmol/L)
Arm/Group | Deferasirox
Number analyzed (Participants) | 57
micromoles per litre (μmol/L)
  Week 8, Deferasirox 20 mg/kg: number analyzed (Participants) | 11
  Week 8, Deferasirox 20 mg/kg | 36.30 [0.0 to 145.0]
  Week 12, Deferasirox 20 mg/kg: number analyzed (Participants) | 8
  Week 12, Deferasirox 20 mg/kg | 66.95 [2.8 to 157.0]
  Week 16, Deferasirox 20 mg/kg: number analyzed (Participants) | 12
  Week 16, Deferasirox 20 mg/kg | 27.75 [0.0 to 200.0]
  Week 8, Deferasirox 30 mg/kg: number analyzed (Participants) | 8
  Week 8, Deferasirox 30 mg/kg | 20.15 [2.2 to 62.1]
  Week 12, Deferasirox 30 mg/kg: number analyzed (Participants) | 9
  Week 12, Deferasirox 30 mg/kg | 34.30 [0.0 to 105.0]
  Week 16, Deferasirox 30 mg/kg: number analyzed (Participants) | 9
  Week 16, Deferasirox 30 mg/kg | 54.50 [0.0 to 146.0]

4. Secondary Outcome: Change From Baseline in Serum Ferritin at Week 16
Description: Ferritin protein stores iron and provides overall iron levels. Higher ferritin in blood showed higher iron content. Fluctuations from normal serum ferritin levels (500 ng/mL) observed at two consecutive visits led to dose adjustment of deferasirox.
Time Frame: Baseline, Week 16 (End of study)
Population: The analysis was performed in the ITT population. The 'n' signifies those subjects evaluable for this measure at specified time points for each group respectively. As per the planned analysis, data was summarized as overall by combining all Arms/Groups.
Measure: Mean (Standard Deviation); unit: Nanogram/mlillilitre
Arm/Group | Deferasirox
Number analyzed (Participants) | 64
Nanogram/mlillilitre
  Age 2 to < 10 years: number analyzed (Participants) | 10
  Age 2 to < 10 years | -198.1 (653.11)
  Age 10 to < 60 years: number analyzed (Participants) | 44
  Age 10 to < 60 years | 38.3 (859.45)
  Age ≥ 60 years: number analyzed (Participants) | 10
  Age ≥ 60 years | -593 (1683.39)

ADVERSE EVENTS:
Time Frame: First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV), up to 16 weeks
Description: The analysis was performed in the Safety Set (SAF) population, defined as all participants who received at least one dose of study medication.
Groups:
- No Meal (Deferasirox With Soft Food): Participants received crushed deferasirox at a minimum starting dose of 20 mg/kg/day added to a soft food with no meal for 12 weeks of assessment period. For participants receiving > 30 mg/kg/ day, a maximum of 40 mg/kg/day was allowed.
- Deferasirox (Overall): Participants were administered daily with deferasirox at a minimum starting dose of 20 mg/kg/day along with different food and liquids consistently for 12 weeks of assessment period. For subjects receiving > 30 mg/kg/day, a maximum of 40 mg/kg/day was allowed.
Arm/Group | Deferasirox (Run-in Phase) | Breakfast (Deferasirox With Soft Food) | Breakfast (Deferasirox With Liquid) | Dinner (Deferasirox With Soft Food) | Dinner (Deferasirox With Liquid) | No Meal (Deferasirox With Liquid) | No Meal (Deferasirox With Soft Food) | Deferasirox (Overall)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/20 | 0/18 | 0/14 | 0/17 | 0/39 | 0/30 | 0/65
Serious Adverse Events (participants affected / at risk) | 5/62 | 5/20 | 0/18 | 1/14 | 1/17 | 6/39 | 0/30 | 15/65
Other Adverse Events (participants affected / at risk) | 30/62 | 10/20 | 6/18 | 6/14 | 6/17 | 18/39 | 9/30 | 52/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (Run-in Phase) (N=62) | Breakfast (Deferasirox With Soft Food) (N=20) | Breakfast (Deferasirox With Liquid) (N=18) | Dinner (Deferasirox With Soft Food) (N=14) | Dinner (Deferasirox With Liquid) (N=17) | No Meal (Deferasirox With Liquid) (N=39) | No Meal (Deferasirox With Soft Food) (N=30) | Deferasirox (Overall) (N=65)
Acute chest syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 3 | 0 | 0 | 0 | 1 | 5 | 0 | 8
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter related complication (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.90% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (Run-in Phase) (N=62) | Breakfast (Deferasirox With Soft Food) (N=20) | Breakfast (Deferasirox With Liquid) (N=18) | Dinner (Deferasirox With Soft Food) (N=14) | Dinner (Deferasirox With Liquid) (N=17) | No Meal (Deferasirox With Liquid) (N=39) | No Meal (Deferasirox With Soft Food) (N=30) | Deferasirox (Overall) (N=65)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 2 | 2 | 0 | 1 | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 3 | 8
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 15 | 1 | 1 | 1 | 0 | 2 | 2 | 20
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 1 | 0 | 2 | 1 | 3 | 0 | 15
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 1 | 0 | 2 | 2 | 10
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Exercise tolerance decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 8
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 7 | 2 | 0 | 3 | 0 | 4 | 1 | 15
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 5 | 1 | 8
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 5
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 5 | 2 | 2 | 0 | 0 | 1 | 1 | 7
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No